CLINICAL TRIAL: NCT06096246
Title: Objective Randomised Blinded Investigation of Cardioversion Versus Ablation for Persistent Atrial Fibrillation (ORBICA-AF)
Brief Title: Investigation of Cardioversion Versus Therapeutic Ablation for Persistent AF (ORBICA-AF)
Acronym: ORBICA-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORBICA-AF
Record Dates: First submitted 2023-09-21; First posted 2023-10-23 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Persistent Atrial Fibrillation; Cardiac Arrhythmia; Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: Randomised, blinded, controlled trial with 2 arms
Who Masked: Participant, Investigator
Masking Description: Patient and physician - blinded randomisation to intervention (DCCV, or Pulmonary Vein Isolation plus DCCV) Once subject participation in the trial is complete, the patient and physician will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: DCCV + PVI (Active Comparator): An implantable loop recorder will be inserted in the pre pectoral area with local anaesthetic at least one week before the randomisation.
  Two femoral sheaths will be inserted at the groin area in all patients on the day of the procedure prior randomisation. This will be utilised as the access route for cardiac catheter insertion for ablation and for phrenic nerve pacing during the procedure.
  DC cardioversion (DCCV) plus Pulmonary Vein Isolation - At the end of pulmonary vein isolation, DCCV is performed (if the patient is still in AF).
  Interventions: Procedure: Pulmonary vein isolation; Procedure: DC Cardioversion; Device: Implantable loop recorder; Procedure: Femoral sheath insertion
- DC cardioversion (DCCV) + Sham procedure (Sham Comparator): An implantable loop recorder will be inserted in the pre-pectoral area with local anaesthetic at least one week before the randomisation.
  Two femoral sheaths will be inserted at the groin area in all patients on the day of the procedure prior randomisation. This will be utilised as the access route for cardiac catheter insertion for intermittent phrenic nerve pacing during the procedure.
  DC Cardioversion and Sham procedure will be performed after randomisation. Intermittent phrenic nerve pacing will be employed for the sham group through the femoral venous sheath using a quadripolar catheter.
  Interventions: Procedure: DC Cardioversion; Device: Implantable loop recorder; Procedure: Femoral sheath insertion

INTERVENTIONS:
Procedure: Pulmonary vein isolation — The catheter ablation (with a CE [Conformité Européenne] marked device) is the key specified technique for performing pulmonary vein isolation in the ablation arm in this trial. This allows the physician electrophysiologist to perform a circumferential ablation around the pulmonary veins to electrically isolate the vein, thus preventing pulmonary vein ectopy from triggering AF.
  Other Names: Catheter ablation
  Arms: Experimental: DCCV + PVI
Procedure: DC Cardioversion — DC cardioversion (DCCV) is used to treat irregular heart rhythms (commonly atrial fibrillation). The procedure involves sedation or anaesthetic and placement of electrodes on the chest. An electrical impulse is passed across the electrodes to return the heart rhythm to normal.
Device: Implantable loop recorder — The Reveal device is inserted in the pre-pectoral position under the skin. This is performed with local anaesthetic and sedation at least a week before the randomisation. The device will provide a continuous recording of the heart rhythm and rate, and will be able to download duration of AF episodes via a home monitoring system to establish the primary endpoint of the study .
  Other Names: Reveal LINQ
Procedure: Femoral sheath insertion — Two femoral sheaths (7Fr) will be inserted using ultrasound guidance under local anaesthetic.

SUMMARY:
The main aim of the research is to investigate whether patients undergoing pulmonary vein isolation with catheter ablation for persistent atrial fibrillation (AF) will have lower rates of AF recurrence than those treated by DC cardioversion without an ablation procedure.

DETAILED DESCRIPTION:
After adequate stroke prevention (e.g. anticoagulation) and rate control, the optimum strategy for patients who continue to be symptomatic with persistent AF has not been established. Cardioversion with antiarrhythmic medication is commonly used as a first-line rhythm control strategy despite very high recurrence rates of index arrhythmia and high serious complications associated with this strategy. Further treatment options, such as catheter ablation or implantation of a pacemaker and ablation of the atrioventricular (AV) node, are considered once AF recurs. The benefits of first-line ablation in patients presenting with persistent AF have not been tested. Investigators seek to perform a blinded, randomised trial comparing an electrical cardioversion-led strategy with a pulmonary-vein isolation strategy for the treatment of persistent atrial fibrillation. No blinded randomised controlled trial comparing early-ablation strategies to cardioversion-led strategies has been performed. The rationale for blinding where possible in clinical trials is well established. The recently published ORBITA trial performed a blinded, multicentre randomised trial of percutaneous coronary intervention (PCI) in stable angina compared to a placebo procedure. This trial demonstrated that the efficacy of invasive procedures can be assessed with a placebo procedure and that this type of trial remains necessary. Knowledge of treatment assignment influences physician behaviour, drug recommendations and encourages bias in outcome reporting. The treatment effect size and the effects of confounding factors will be exaggerated and thus limit the interpretation of the true patient-experienced outcomes of either strategy. In a comparison of surgical procedures, a sham control arm represents the gold standard of blinding. A systematic review of placebo-controlled surgical trials found no evidence of harm to participants assigned to the placebo group. For a procedure whose primary purpose is to give sustained symptomatic relief, definitive quantification of the true placebo-controlled effect size of AF ablation is necessary. There is a need to clarify the relationship between patient-reported symptoms and the arrhythmia itself. Patient-reported symptoms may not always be related to the severity of the arrhythmia or quality of life. No bias-resistant blinded, randomised, trial has yet been performed seeking to measure the benefits of AF ablation in persistent AF. The investigators of this trial have achieved successful recruitment and concluded the pilot phase (ORBITA AF trial; ClinicalTrials.gov Identifier: NCT03907982) with the goal of assessing feasibility and optimizing the study protocol prior to conducting a larger trial. The positive outcomes of the pilot phase have paved the way for this larger follow-on trial.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Age 18-85 years
* Persistent AF (atrial fibrillation lasting > 7days) of total continuous duration <2 years as documented in medical notes.
* Patients being considered for cardioversion.

Exclusion Criteria:

* Creatinine clearance (eGFR) < 30mls/min
* Contraindication or unable to take anticoagulation
* Uncontrolled hypertension
* Contraindication for catheter ablation
* BMI > 40
* Patients in Persistent AF who have had more than one previous cardioversion.
* Established diagnosis of Hypertrophic cardiomyopathy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2027-07-26 (Estimated); Study Completion 2027-12-05 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Persistent AF (AF episode lasting > 7 days) or left atrial ablation/ DC Cardioversion for atrial arrhythmia after 6 weeks of blanking period. | Within 12 months following the procedure
  Rates of recurrence of arrhythmia and data on episodes of Atrial Fibrillation (rate, duration) will be provided by the loop recorder, and downloaded via a home monitoring system [ rhythm on ILR ECG]
A change in the burden of AF, as measured by continuous monitoring through ILR (Implantable loop recorder) at 3 months | 3 months post randomisation
  Percentage time the patient is in AF as measured by the ILR device (in percentage) compared to pre-randomisation

SECONDARY OUTCOMES:
Death | Within 12 months of study index procedure.
  Death of the patient
Rates of Subject Hospital re-admission | Within 12 months of study index procedure.
  Rates of admission of the subject back to hospital following the initial treatment for AF
Procedural complications | Up to 7 days post procedure
  Assessment of rates of events that are considered procedural complications during the DCCV +/- Pulmonary Vein isolation (PVI) procedure
Bleeding events | Within 7 days of the index procedure
  Rates of bleeding in subjects following the study DCCV +/- pulmonary vein isolation (PVI) procedures
Rates of Repeat procedures | within 12 months following the procedure
  Requirement for repeat procedures following the initial DCCV +/- pulmonary vein isolation (PVI) procedure for the study
Cardiac function | between baseline and 12 months following the procedure
  Measurement of change in ejection fraction by echocardiogram
Percentage of clinical success of procedure | Within 12 months following the index procedure
  Clinical procedural success as defined by 75% or greater reduction in the number of AF episodes as measured by the insertable cardiac monitoring system (LINQ) device.
Change in quality of life score using in 12 item Short Form health survey (SF12) | Between baseline and 3, 6 and 12 months after procedure
  Assessment of quality of life measures using Short Form Health Survey (SF12) questionnaire, which is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey. The questions are combined, scored, and weighted to create two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Change in quality of life measures using Atrial Fibrillation Effect on QualiTy-of-life(AFEQT) questionnaire | Between baseline and 3, 6 and 12 months after procedure
  Assessment of AF specific symptoms to assess the impact of AF on the subject's quality of life. The responses on the 20-item AFEQT are scored on a 1 to 7 Likert scale. Overall and subscale scores range from 0 to 100. A score of 0 corresponds to complete disability, while a score of 100 describes the highest level of QoL
Measuring Blinding index | Day 0 (within 24 hours post randomisation) and 3 months
  Assessing the maintenance of blinding measured by Blinding index in both study participant and blinded medical staff.
Measuring AF Burden | At 3, 6 and 12 months follow up
  Percentage time the patient is in AF as measured by the ILR (Implantable loop recorder) device compared to pre-randomisation
The occurrence of atrial tachyarrhythmias | Within 12 months following the index procedure
  Assessment of the occurence of other atrial tachyarrhythmia (Atrial flutter or Atrial tachycardia) in the continuous monitoring
Symptomatic Atrial fibrillation/Atrial tachycardia episodes | At 3, 6, 12 months follow up
  Number of symptomatic AF/AT triggered/reported by patients correlating to true episodes in the continuous monitoring.
Antiarrhythmic drug use | Between baseline and 12months after procedure
  Assessment of the use of antiarrhythmic drugs (combined data collected on duration , dose and frequency of drug use) prior to and after the DCCV +/- PVI procedure
Composite adverse events | 12 months
  Assessment of rates of adverse events during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schilling, FRCP MD, Study Chair — Barts & The London NHS Trust; Malcolm Finlay, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Barts Heart Centre, London, United Kingdom

REFERENCES:
- [Result] Wartolowska K, Judge A, Hopewell S, Collins GS, Dean BJ, Rombach I, Brindley D, Savulescu J, Beard DJ, Carr AJ. Use of placebo controls in the evaluation of surgery: systematic review. BMJ. 2014 May 21;348:g3253. doi: 10.1136/bmj.g3253. PMID 24850821
- [Result] Redberg RF. Sham controls in medical device trials. N Engl J Med. 2014 Sep 4;371(10):892-3. doi: 10.1056/NEJMp1406388. No abstract available. PMID 25184861
- [Result] Miller FG, Kaptchuk TJ. Sham procedures and the ethics of clinical trials. J R Soc Med. 2004 Dec;97(12):576-8. doi: 10.1177/014107680409701205. No abstract available. PMID 15574854
- [Result] Jones C, Pollit V, Fitzmaurice D, Cowan C; Guideline Development Group. The management of atrial fibrillation: summary of updated NICE guidance. BMJ. 2014 Jun 19;348:g3655. doi: 10.1136/bmj.g3655. No abstract available. PMID 24948694
- [Result] Brim RL, Miller FG. The potential benefit of the placebo effect in sham-controlled trials: implications for risk-benefit assessments and informed consent. J Med Ethics. 2013 Nov;39(11):703-7. doi: 10.1136/medethics-2012-101045. Epub 2012 Dec 13. PMID 23239742
- [Result] Al-Lamee R, Thompson D, Dehbi HM, Sen S, Tang K, Davies J, Keeble T, Mielewczik M, Kaprielian R, Malik IS, Nijjer SS, Petraco R, Cook C, Ahmad Y, Howard J, Baker C, Sharp A, Gerber R, Talwar S, Assomull R, Mayet J, Wensel R, Collier D, Shun-Shin M, Thom SA, Davies JE, Francis DP; ORBITA investigators. Percutaneous coronary intervention in stable angina (ORBITA): a double-blind, randomised controlled trial. Lancet. 2018 Jan 6;391(10115):31-40. doi: 10.1016/S0140-6736(17)32714-9. Epub 2017 Nov 2. PMID 29103656
- [Result] Bang H, Ni L, Davis CE. Assessment of blinding in clinical trials. Control Clin Trials. 2004 Apr;25(2):143-56. doi: 10.1016/j.cct.2003.10.016. PMID 15020033